CLINICAL TRIAL: NCT02708446
Title: A Randomized Controlled Trial to Compare Sublingual and Buccal Misoprostol Regimens After Mifepristone for Termination of Pregnancy 13 - 21 Weeks From Last Menstrual Period (LMP)
Brief Title: A Comparison of Sublingual and Buccal Misoprostol Regimens After Mifepristone for Mid-trimester Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gynuity Health Projects (Other)
Collaborators: La Rabta Maternity Hospital (Unknown); Republican Institute of RH, Perinatology, and Ob/Gyn (Unknown); Kathmandu Medical College and Teaching Hospital (Other); Clinic No. 2 of Tashkent Medical Academy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1013
Record Dates: First submitted 2016-02-10; First posted 2016-03-15 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Legally Induced Abortion Without Mention of Complication
Keywords: Second Trimester; Abortion; Misoprostol; Sublingual; Buccal
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sublingual misoprostol (Active Comparator): 200mg mifepristone + 400mcg sublingual misoprostol q3h
  Interventions: Drug: Mifepristone; Drug: Sublingual misoprostol
- Buccal misoprostol (Active Comparator): 200mg mifepristone + 400mcg buccal misoprostol q3h
  Interventions: Drug: Mifepristone; Drug: Buccal misoprostol

INTERVENTIONS:
Drug: Mifepristone — 200mg oral mifepristone to both study arms
  Other Names: miropristone; Mifeprex; Mifegyne
Drug: Buccal misoprostol — doses of buccal misoprostol every 3 hours beginning 24 hours after mifepristone
  Other Names: cytotec
  Arms: Buccal misoprostol
Drug: Sublingual misoprostol — doses of sublingual misoprostol every 3 hours beginning 24 hours after mifepristone
  Other Names: cytotec
  Arms: Sublingual misoprostol

SUMMARY:
The primary goal of this study is to directly compare repeat doses of sublingual and buccal routes of 400 mcg misoprostol following mifepristone for second trimester abortion in order to determine if sublingual route confers an advantage with respect to efficacy and median time to complete abortion.

DETAILED DESCRIPTION:
Eligible women 13-21 weeks gestation who give informed consent will be randomized to receive buccal or sublingual misoprostol. Participants will take 200mg mifepristone and return to the hospital 24 hours later to begin induction with misoprostol. 400mcg misoprostol will be given every 3 hours until the expulsion of the fetus and placenta.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria to obtain abortion
* Present with closed cervical os and no vaginal bleeding
* Live fetus at time of presentation for service
* Have no contraindications to study procedures, according to provider
* Be able to consent to procedure, either by reading consent document or by having consent document read to her
* Be willing to follow study procedures

Exclusion Criteria:

* Known previous transmural uterine incision
* Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
* Any contraindications to vaginal delivery
* Presentation in active labor (defined as moderate to severe contractions every 10 minutes or less)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rate of successful abortion by 24 hours | 24 hours following the start of misoprostol
  Defined as complete evacuation of uterus at 24 hours following start of misoprostol, using study drugs without recourse to any additional intervention.
Rate of successful abortion by 48 hours | 48hours following the start of misoprostol
  Defined as complete evacuation of uterus at 48 hours following start of misoprostol, using study drugs without recourse to any additional intervention.

SECONDARY OUTCOMES:
Median time from first dose of misoprostol to complete expulsion of complete expulsion (provider diagnosis of complete expulsion of fetus and placenta). | 48 hours
Percentage of patients requiring provision of additional interventions. | from first drug dose to complete expulsion as documented on study forms, up to 72 hours
Total number of doses of misoprostol. | from first drug dose to complete expulsion as documented on study forms, up to 72 hours
Rates of heavy bleeding, uterine rupture, or infection requiring additional treatment | 1 month
Pain scale (1-7) as reported by women on questionnaire | from first drug dose to complete expulsion as documented on study forms, up to 72 hours
Women's acceptability of the assigned method based on 5 point acceptability scale in questionnaire | from first drug dose to complete expulsion as documented on study forms, up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (4):
- b. Republican Institute of Reproductive Health, Perinatology, Obstetrics and Gynecology (RIRHPOG), Yerevan, Armenia
- Kathmandu Medical College, Kathmandu, Nepal
- La Rabta Maternity Hospital, Tunis, Tunisia
- Clinic No. 2, Tashkent Medical Academy, Tashkent, Uzbekistan